CLINICAL TRIAL: NCT01585792
Title: Double Blind Comparative Study of TAK-875
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: TAK-875/CPH-030; U1111-1129-7907 (Registry Identifier: WHO); JapicCTI-121816 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Diabetic Patients
MeSH Terms: interventions — TAK-875; glimepiride

ARMS (4):
- TAK-875 25 mg (Experimental)
  Interventions: Drug: TAK-875
- TAK-875 50 mg (Experimental)
  Interventions: Drug: TAK-875
- Glimepiride (Active Comparator)
  Interventions: Drug: Glimepiride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-875
  Arms: TAK-875 25 mg
Drug: TAK-875
  Arms: TAK-875 50 mg
Drug: Glimepiride
  Arms: Glimepiride
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of treatment with TAK-875 in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* The participant is an outpatient.
* The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

* The participant has any serious cardiac disease, serious cerebrovascular disorder, or any serious pancreatic or hematological disease.
* The participant is considered ineligible for the study for any other reason by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 4 weeks
  Blood glucose

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Fukuoka, Fukuoka
  - Sumida-ku, Tokyo